CLINICAL TRIAL: NCT02266576
Title: A Patient-Centered Strategy for Improving Diabetes Prevention in Urban American Indians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: San Jose State University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Randall Stafford, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SU-30015; PCORI-PCORIAD-1306-02172 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Diabetes Prevention Program (DPP) (Active Comparator): Participants receive Standard DPP over the course of 20 weeks.
  Interventions: Behavioral: Standard DPP
- Enhanced DPP (Experimental): Participants receive Standard DPP plus Enhanced DPP over the course of 20 weeks.
  Interventions: Behavioral: Standard DPP; Behavioral: Enhanced DPP

INTERVENTIONS:
Behavioral: Standard DPP — The Standard Diabetes Prevention Program (DPP) delivered by the San Jose State Timpany Center is the Group Lifestyle Balance™ DPP, which has previously been tailored for urban American Indians and Alaska Natives by the Indian Health Service. Standard DPP components consist of 16 group classes, 4 visits with a lifestyle coach and access to a therapeutic swimming pool and gym.
Behavioral: Enhanced DPP — Enhanced DPP components consist of access to a mental health counselor, active referrals to mental health services, and traditional healing workshops such as the use of talking circles, a modified photo voice and digital storytelling to address specific psychosocial issues that are a result of historical trauma, stress, and grief.
  Arms: Enhanced DPP

SUMMARY:
The goal of the proposed research is to identify effective patient-centered strategies to prevent diabetes in high-risk populations in real world settings. The investigators will accomplish this by conducting a randomized controlled trial comparing an enhanced Diabetes Prevention Program addressing psychosocial stressors to a standard version in a high-risk population of urban American Indian and Alaska Native people within a primary care setting.

DETAILED DESCRIPTION:
The goal of the proposed research is to identify effective patient-centered strategies to prevent diabetes in high-risk populations in real world settings. The investigators will accomplish this by conducting a randomized controlled trial comparing an enhanced Diabetes Prevention Program addressing psychosocial stressors to a standard version in a high-risk population of urban American Indian and Alaska Native peoples within a primary care setting. Diabetes is disproportionately prevalent among low-socioeconomic status and racial/ethnic minority populations in the US. The high prevalence of psychosocial stressors such as depression, discrimination, and exposure to trauma among these populations contributes to the high prevalence of diabetes and interferes with successful completion of lifestyle interventions. The investigators hypothesize that a DPP that directly addresses these psychosocial stressors will be superior to the standard DPP in addressing this disparity in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Urban of Indigenous Ancestry from the Americas (North, Central and South America)
* Men and women
* BMI Between 30-55
* Not diagnosed with Type II Diabetes
* At least one of the following criterion

  1. Triglycerides: 150mg/dL or higher
  2. Reduced HDL: <40mg/dL (men); <50mg/dL (women)
  3. Blood pressure: >130/80 or current treatment with antihypertensives
  4. Fasting glucose: >100mg/dL

Exclusion Criteria:

* Significant medical comorbidities, including uncontrolled metabolic disorders (e.g., thyroid, diabetes, renal, liver), unstable heart disease, heart failure, and ongoing substance abuse;
* On greater than 10 prescription medications.
* Psychiatric disorders requiring atypical antipsychotics or multiple medications;
* Inappropriate for moderate exercise according to the Revised Physical Activity Readiness Questionnaire;
* Pregnant, planning to become pregnant, or lactating;
* Family household member already enrolled in the study;
* Already enrolled or planning to enroll in a clinical trial that would limit full participation in the study;
* Resident of a long term care facility;
* Lack of spoken English by patient or a household member > 18 y who can serve as interpreter;
* Plans to move during the study period (9 months post-randomization);
* Investigator discretion for clinical safety or adherence reasons (e.g., unstable housing, chronic pain).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall S Stafford, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Timpany Center of San Jose State University, San Jose, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Background] Rosas LG, Vasquez JJ, Naderi R, Jeffery N, Hedlin H, Qin F, LaFromboise T, Megginson N, Pasqua C, Flores O, McClinton-Brown R, Evans J, Stafford RS. Development and evaluation of an enhanced diabetes prevention program with psychosocial support for urban American Indians and Alaska natives: A randomized controlled trial. Contemp Clin Trials. 2016 Sep;50:28-36. doi: 10.1016/j.cct.2016.06.015. Epub 2016 Jul 2. PMID 27381232
- [Derived] Rosas LG, Vasquez JJ, Hedlin HK, Qin FF, Lv N, Xiao L, Kendrick A, Atencio D, Stafford RS. Comparing enhanced versus standard Diabetes Prevention Program among indigenous adults in an urban setting: a randomized controlled trial. BMC Public Health. 2020 Jan 30;20(1):139. doi: 10.1186/s12889-020-8250-7. PMID 32000738

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Diabetes Prevention Program (DPP): Participants receive Standard DPP (Group Lifestyle Balance™ DPP delivered by the San Jose State Timpany Center) over the course of 20 weeks. Standard DPP components consist of 16 group classes, 4 visits with a lifestyle coach and access to a therapeutic swimming pool and gym.
- Enhanced DPP: Participants receive Enhanced DPP over the course of 20 weeks. Enhanced DPP components consist of Standard DPP components, plus access to a mental health counselor, active referrals to mental health services, and traditional healing workshops such as the use of talking circles, a modified photo voice and digital storytelling to address specific psychosocial issues that are a result of historical trauma, stress, and grief.
Period: Overall Study
Arm/Group | Standard Diabetes Prevention Program (DPP) | Enhanced DPP
Started | 102 | 105
Completed | 85 | 90
Not Completed | 17 | 15

BASELINE CHARACTERISTICS:
Groups:
- Standard DPP: Participants receive Standard DPP over the course of 20 weeks. Standard DPP components consist of 16 group classes, 4 visits with a lifestyle coach and access to a therapeutic swimming pool and gym.
- Enhanced DPP: Participants receive Enhanced DPP over the course of 20 weeks. Enhanced DPP components consist of Standard DPP components, plus access to a mental health counselor, active referrals to mental health services, and traditional healing workshops, such as the use of talking circles, and modified photo voice and digital storytelling to address specific psychosocial issues that are a result of historical trauma, stress, and grief.
- Total: Total of all reporting groups
Arm/Group | Standard DPP | Enhanced DPP | Total
Number analyzed (Participants) | 102 | 105 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.8) | 52.1 (13.8) | 52.0 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 83 | 163
  Male | 22 | 22 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 56 | 112
  Not Hispanic or Latino | 46 | 49 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 102 | 105 | 207
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2]
  Men | 35.5 (4.7) | 39.5 (7.8) | 37.5 (6.6)
  Women | 37.1 (5.8) | 37.2 (6.2) | 37.2 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Mass Index (BMI) Through Month 12
Description: BMI is measured as weight in kg divided by the square of height in meters.
Time Frame: Change through month 12, with assessments at baseline, 6 months, and 12 months
Population: One participant from each group was excluded at baseline due to safety concerns; participants with available data at subsequent time points were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Standard DPP | Enhanced DPP
Number analyzed (Participants) | 101 | 104
kg/m^2
  Baseline | 37.0 [35.63 to 38.37] | 37.8 [36.43 to 39.17]
  Change from baseline to month 6: number analyzed (Participants) | 79 | 78
  Change from baseline to month 6 | -.7 [-1 to -.4] | -.3 [-0.7 to -.02]
  Change in baseline to month 12: number analyzed (Participants) | 85 | 90
  Change in baseline to month 12 | -.5 [-1 to -.1] | -.3 [-.7 to .2]
Statistical Analysis 1: Comparison: Standard DPP vs Enhanced DPP; Baseline vs month 6; Test type: Other; p = 0.04, Regression, Linear — The linear regression model was used, adjusted for within cohort correlation, within participant correlation, and gender
Statistical Analysis 2: Comparison: Standard DPP vs Enhanced DPP; Baseline vs month 12; Test type: Other; p = 0.02, Regression, Linear; The linear regression model was used, adjusted for within cohort correlation, within participant correlation, and gender

2. Primary Outcome: Change From Baseline in the Quality of Life Short Form Survey (SF-12)
Description: SF-12 scale is a generic, multipurpose short-form survey with 12 questions selected from the SF-36 Health Survey to evaluate overall health-related quality of life. Answers are combined, scored and weighted into mental and physical functioning component scales. The scores for each scale range from 0 to 100. A higher value indicates a better quality of life of the patient.
Time Frame: Change through month 12, with assessments at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard DPP | Enhanced DPP
Number analyzed (Participants) | 101 | 104
score on a scale
  Physical-baseline | 41.5 [38.95 to 44.05] | 40.2 [37.65 to 42.75]
  Physical-change from baseline at month 6: number analyzed (Participants) | 79 | 78
  Physical-change from baseline at month 6 | 3.0 [.9 to 5.1] | 3.1 [1 to 5.2]
  Physical-change from baseline at month 12: number analyzed (Participants) | 85 | 90
  Physical-change from baseline at month 12 | 2.2 [-.1 to 4.5] | 2.9 [.7 to 5.2]
  Mental-baseline | 47.1 [44.75 to 49.45] | 48 [45.65 to 50.35]
  Mental-change from baseline at month 6: number analyzed (Participants) | 79 | 78
  Mental-change from baseline at month 6 | 1.5 [-1.1 to 4.2] | 1.7 [-1.0 to 4.3]
  Mental-change from baseline at month 12: number analyzed (Participants) | 85 | 90
  Mental-change from baseline at month 12 | 2 [-.7 to 4.7] | .3 [-2.4 to 3]
Statistical Analysis 1: Comparison: Standard DPP vs Enhanced DPP; Baseline vs month 6 in physical component score; Test type: Other; p = 0.004, Regression, Linear; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Standard DPP vs Enhanced DPP; Baseline vs month 12 in physical component score; Test type: Other; p = 0.01, Regression, Linear; [statistical method as in outcome 1, analysis 2]

3. Secondary Outcome: Change From Baseline in Food Frequency Questionnaire (FFQ) Score as a Measure of Healthy and Unhealthy Diet Choices
Description: The FFQ modified to incorporate culturally-relevant food choices (e.g. corn tortillas and frybread) was used. Food items were scored on a scale of 1 to 6 (6 corresponding to the greatest frequency of consumption), and categorized as "healthy," "unhealthy," and "undetermined" based on classifications previously determined by Teuful-Shone et al. "Healthy" foods were those recommended for increased intake (e.g. green leafy salad). "Unhealthy" foods were recommended for decreased intake (e.g. soft drinks), and all remaining foods were "undetermined." Healthy and unhealthy food scores (but not undetermined) were collected for this outcome measure. Scores were summed for a total score. Healthy food choices (6 questions) score range 3-36 (higher scores mean healthier diet). Unhealthy food choices (13 questions) score range: 13-78 (lower scores mean healthier diet).
Time Frame: Change through month 12, with assessments at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard DPP | Enhanced DPP
Number analyzed (Participants) | 101 | 104
score on a scale
  Healthy (baseline) | 22.6 [21.62 to 23.58] | 22.8 [21.82 to 23.78]
  Healthy (month 6): number analyzed (Participants) | 79 | 78
  Healthy (month 6) | -.6 [-1.7 to .5] | .4 [-0.7 to 1.5]
  Healthy (month 12): number analyzed (Participants) | 85 | 90
  Healthy (month 12) | 0.4 [-0.9 to 1.7] | -0.4 [-1.6 to 0.9]
  Unhealthy (baseline) | 37.9 [35.94 to 39.86] | 35.4 [33.44 to 37.36]
  Unhealthy (month 6): number analyzed (Participants) | 79 | 78
  Unhealthy (month 6) | -4.6 [-6.5 to -2.8] | -2.51 [-4.4 to -0.6]
  Unhealthy (month 12): number analyzed (Participants) | 85 | 90
  Unhealthy (month 12) | -4.6 [-6.8 to -2.5] | -0.7 [-2.9 to 1.4]

4. Secondary Outcome: Change From Baseline in Physical Activity Measured in Metabolic Equivalents (MET) Per Week
Description: MET is a term used to represent the intensity of exercise. A MET is the ratio of the rate of energy expended during an activity to the rate of energy expended at rest. At least 1000 MET minutes per week are needed to lower the risk of disease.
  * 1 minute of light-intensity activities = 1.1 MET to 2.9 METs
  * 1 minute of moderate-intensity activities = 3.0 to 5.9 METs
  * 1 minute of vigorous-intensity activities = 6.0 METs or more
Time Frame: Change through month 12, with assessments at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: MET minutes per week
Arm/Group | Standard DPP | Enhanced DPP
Number analyzed (Participants) | 101 | 104
MET minutes per week
  Baseline | 1389.1 [1095.69 to 1682.51] | 1541 [1246.01 to 1835.19]
  Change from baseline at month 6: number analyzed (Participants) | 79 | 78
  Change from baseline at month 6 | -94.3 [-386.2 to 197.6] | -23.5 [-314.8 to 267.8]
  Change from baseline at month 12: number analyzed (Participants) | 85 | 90
  Change from baseline at month 12 | 144.6 [-207.6 to 496.8] | -241.6 [-591.9 to 108.7]

5. Secondary Outcome: Change From Baseline in the Center for Epidemiologic Studies - Depression Scale (CES-D) as a Measure of Mental Health Symptoms
Description: The CES-D (Radloff, 1977) is a 20-item, self-report scale designed to assess the presence and severity of depressive symptoms over the past week. The total range is 0-80, with higher scores reflecting more severe depression symptoms.
Time Frame: Change through month 12, with assessments at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard DPP | Enhanced DPP
Number analyzed (Participants) | 101 | 104
score on a scale
  Baseline | 13.9 [11.55 to 16.25] | 12.2 [10.04 to 14.36]
  Change from baseline at month 6: number analyzed (Participants) | 79 | 78
  Change from baseline at month 6 | -2.3 [-4.6 to -0.1] | 0.04 [-2.2 to 2.3]
  Change from baseline at month 12: number analyzed (Participants) | 85 | 90
  Change from baseline at month 12 | -1.2 [-3.8 to 1.5] | -0.1 [-2.7 to 2.6]

6. Secondary Outcome: Change From Baseline in Empowerment
Description: The Growth and Empowerment Measure (GEM) was developed to measure change in dimensions of empowerment as defined and described by Aboriginal Australians who participated in the Family Well Being programme. The GEM has two components. The 14-item Emotional Empowerment Scale has a range of 12-60, with higher scores corresponding to more ability to feel and show the signs of empowerment . The 12-item Scenarios scale has a range of 12-84, with higher scores corresponding to better emotional empowerment in different scenarios.
Time Frame: Change through month 12, with assessments at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard DPP | Enhanced DPP
Number analyzed (Participants) | 101 | 104
score on a scale
  Emotional empowerment (baseline) | 46.2 [44.04 to 48.36] | 47.1 [44.94 to 49.26]
  Change from baseline emotional empowerment (mo 6): number analyzed (Participants) | 79 | 78
  Change from baseline emotional empowerment (mo 6) | 0.2 [-2 to 2.5] | -0.4 [-2.7 to 1.9]
  Change from baseline emotional empowerment (mo12): number analyzed (Participants) | 85 | 90
  Change from baseline emotional empowerment (mo12) | -0.3 [-2.7 to 2] | 0.9 [-1.5 to 3.2]
  Scenarios (baseline) | 59.9 [56.37 to 63.43] | 57.1 [53.77 to 60.43]
  Change from baseline scenarios (month 6): number analyzed (Participants) | 79 | 78
  Change from baseline scenarios (month 6) | -2.3 [-5.6 to 1] | -1.9 [-5.1 to 1.3]
  Change from baseline scenarios (month 12): number analyzed (Participants) | 85 | 90
  Change from baseline scenarios (month 12) | 0.2 [-3.1 to 3.5] | -2.1 [-5.3 to 1.2]

7. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Blood pressure readings are expressed in millimeters of mercury. This unit is abbreviated as mm Hg. A normal reading would be any blood pressure below 120/80 mm Hg and above 90/60 mm Hg in an adult.
Time Frame: Baseline, 6 months and 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: Blood pressure readings are expressed in millimeters of mercury (mmHg). A normal reading would be any blood pressure below 120/80 mm Hg and above 90/60 mm Hg in an adult.
Time Frame: Baseline, 6 months and 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Fasting Blood Glucose
Description: Performed via fasting participant finger stick with Alere Cholestech LDX POS device.
Time Frame: Baseline, 6 months and 12 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Symptoms of Historical Trauma
Description: By patient report using a modified version of the Indigenous People's Survey
Time Frame: Baseline, 6 months and 12 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Waist Circumference
Description: In centimeters, measured by trained assessor using standard protocol
Time Frame: Baseline, 6 months and 12 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Lipid Bioassays
Description: LDL-cholesterol, HDL-cholesterol, and Triglycerides; performed via fasting participant finger stick with Alere Cholestech LDX POS device
Time Frame: Baseline, 6 months and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Standard DPP | Enhanced DPP
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/105
Other Adverse Events (participants affected / at risk) | 0/102 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon approval of community advisory board.

DOCUMENTS (2):
  • Study Protocol (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT02266576/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT02266576/SAP_001.pdf